CLINICAL TRIAL: NCT07208032
Title: Efficacy and Safety of STP Pulsed Radiofrequency Versus Regular Pulsed Radiofrequency for Treatment of Post Herpetic Neuralgia
Brief Title: Pulsed Radiofrequency in Post Herptic Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Elhalwagy, Lecturer of anaesthesia and pain management, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-25-2-7PD
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-02

CONDITIONS: Postherpetic Neuralgia (PHN)
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irregular pulsed Radiofrequency treatment (STP) (Active Comparator)
  Interventions: Procedure: Irregular Pulsed Radiofrequency (STP)
- Regular pulsed Radiofrequency treatment (Active Comparator)
  Interventions: Procedure: regular pulsed Radiofrequency

INTERVENTIONS:
Procedure: Irregular Pulsed Radiofrequency (STP) — Flouroscopic guided irregular pulsed Radiofrequency (STP) for dorsal root ganglion
  Arms: Irregular pulsed Radiofrequency treatment (STP)
Procedure: regular pulsed Radiofrequency — Fluoroscopic guided regular pulsed Radiofrequency for the dorsal root ganglion
  Arms: Regular pulsed Radiofrequency treatment

SUMMARY:
Comparing between regular pulsed Radiofrequency and irregular pulsed Radiofrequency for treatment of postherpetic neuralgia

ELIGIBILITY:
Inclusion Criteria:

Patients with Herps Zoster neuralgia lasting more than one month Neck thoracic lumbar ganglion involvement Refractory to conventional therapy

Exclusion Criteria:

Infection ,tumour at the puncture site Severe cardiovascular or cerebrovascular disease Liver, kidney dysfunction Abnormal coagulation Uncontrolled DM Psychatric diseases Patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain level by Numerical Rating Scale | One day , One week , One month ,Three months postprocedure.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Medical research ethics committee, Sohag, Sohag Governorate
  - Medical research ethics committee, Sohag

IPD SHARING:
Plan to Share IPD: No